CLINICAL TRIAL: NCT04753541
Title: Untersuchung Des Einflusses Von Genetischem Risiko Auf Den Erfolg Einer Katheterablation Bei Paroxysmalem Und Persistierendem Vorhofflimmern
Brief Title: The Influence of Genetic Predisposition on Outcome After Catheter Ablation of Atrial Fibrillation.
Acronym: AF GEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: 304/20 S-KH
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 ml EDTA-blood routine samples taken will be analysed for risk allele loci associated with atrial fibrillation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — this is not an interventional study

SUMMARY:
Catheter ablation is an established standard therapy in interventional treatment of atrial fibrillation.The trial investigates the influence of genetic risk for the recurrence of atrial fibrillation after catheter ablation.

DETAILED DESCRIPTION:
Catheter ablation is an established standard therapy in interventional treatment of atrial fibrillation. electric isolation of the pulmonary veins, from which atrial fibrillation is originating in most patients, is cornerstone of all atrial fibrillation patients.

The most common cause for AF recurrence is still incomplete isolation of the pulmonary veins, on the other hand, only 80% of paroxysmal and 60 % of persistent patients can successfully be cured from atrial fibrillation (despite of isolated pulmonary veins after multiple ablation procedures).

By now, non-procedure related predictive risk factors, resulting in recurrence of atrial fibrillation after catheter ablation, are only partially identified, such as obesity, hypertension and sleep apnea.

In the past year several genetic risk alleles were identified, which are associated with atrial fibrillation. By now the relation between genetic risk, which is determined for every patient by its specific genotype and the outcome of catheter ablation in paroxysmal and persistent atrial fibrillation has not yet been investigated.

The aim is to investigate the influence of genetic risk for the recurrence of atrial fibrillation after catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for primary ablation due to paroxysmale or persistent atrial fibrillation
* written informed consent

Exclusion Criteria:

* patients under 18 years of age or patients not able to give informed consent
* prior left atrial ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients planned for primary ablation due to paroxysmale or persistent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Influence of genetic risk on atrial fibrillation | 10ml blood sample taken at baseline visit (routine blood sample)
  Analysation of the influence of genetic risk on the probability of recurrence of atrial fibrillation after catheter ablation

CONTACTS AND LOCATIONS:
Overall Officials: Bourier Felix, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany

IPD SHARING:
Plan to Share IPD: No